CLINICAL TRIAL: NCT06763562
Title: The Impact of Different Food Orders on Blood Glucose and Fuel Use At Rest
Brief Title: Food Orders on Blood Glucose and Fuel Use At Rest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Associate Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-163
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Glucose Metabolism Disorders; Hunger; Fat Burn
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrate-first meal (Experimental)
  Interventions: Other: Carbohydrate-first meal
- Carbohydrate-last meal (Experimental)
  Interventions: Other: Carbohydrate-last meal

INTERVENTIONS:
Other: Carbohydrate-first meal — Rice eaten first (150 grams), followed by edamame (150 grams) and butter (10 grams)
  Arms: Carbohydrate-first meal
Other: Carbohydrate-last meal — Edamame (150 grams) and butter (10 grams) eaten first, followed by rice (150 grams)
  Arms: Carbohydrate-last meal

SUMMARY:
Consuming a carbohydrate-rich food as the final food in a meal, as compared to the first food in a meal, has been shown to reduce blood glucose levels after eating in both diabetes patients and in healthy controls. However, gaps remain in the literature in this area of research, and currently little is known about how substrate (fuel) use is impacted by altering food order. In addition, most studies to date have used a mix of meat and plant foods, while little research has focused exclusively on vegetarian foods. This randomized experiment will examine how altering the order of foods eaten in a vegetarian meal impacts blood glucose and fuel utilization at rest.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Free from any allergy or condition that precluding consumption of edamame, butter, and rice
* Not currently pregnant
* Free of any medical conditions requiring the use of insulin
* Have no history of bariatric surgery
* Have no implanted electrical devices such as a pacemaker

Exclusion Criteria:

* Younger than 18 and older than 70 years old
* Having an allergy or condition that precludes consumption of edamame, butter, and rice
* Currently pregnant
* Any medical conditions requiring the use of insulin
* A history of bariatric surgery
* Having an implanted electrical device such as a pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory exchange ratio | 90 minutes (baseline/premeal and at 30, 60, and 90 minutes postmeal)
  Ratio of carbon dioxide production and oxygen consumption for determination of fuel use

SECONDARY OUTCOMES:
Fat use | 90 minutes (baseline/premeal and at 30, 60, and 90 minutes postmeal)
  Fat utilization will be estimated from respiratory gas exchange
Carbohydrate use | 90 minutes (baseline/premeal and at 30, 60, and 90 minutes postmeal)
  Carbohydrate utilization will be estimated from respiratory gas exchange
Blood glucose | 90 minutes (baseline/premeal and 30, 60, and 90 minutes postmeal)
  Blood glucose will be measured with fingerstick samples and a portable glucometer
Hunger-satiety perceptions | 90 minutes (baseline/premeal and 30, 60, and 90 minutes postmeal)
  Hunger, appetite, satiety, and fullness on a 0-10 Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Old Dominion University Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared as supplementary material associated with the published peer-reviewed publication or through a publicly available repository (depending on the journal's preference).
Time Frame: Data will become available once the associated article is officially published. The data will be made available indefinitely.